CLINICAL TRIAL: NCT07292662
Title: TAP Block Versus ESP Block in Patients Undergoing Elective Cesarean Section: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6334/AO/25
Record Dates: First submitted 2025-09-12; First posted 2025-12-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Delivery; Regional Anesthesia Block
Keywords: ESP block; TAP block; cesarean section

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessor and investigator will be blind of the procedure as each patient will be associated with an unique ID.
  Patients and patient care provider could not be blind given the nature of the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Active Comparator): Patients will undergo preoperative bilateral TAP block with ropivacaine 0.375% 20 mL per side (total 40 mL)
  Interventions: Procedure: TAP block
- ESP block (Experimental): Patients will undergo preoperative bilateral ESP block with ropivacaine 0.375% 20 mL per side (total 40 mL)
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: TAP block — TAP block will be performed with with ropivacaine 0.375% 20 mL per side (total 40 mL)
  Arms: TAP block
Procedure: ESP block — ESP block will be performed with ropivacaine 0.375% 20 mL per side (total 40 mL)
  Arms: ESP block

SUMMARY:
This study is comparing two types of pain relief techniques-TAP block and ESP block-for women having an elective cesarean section. Both techniques involve injecting local anesthetic under ultrasound guidance to numb nerves and reduce pain after surgery. The TAP block mainly relieves pain in the abdominal wall, while the ESP block may reduce both abdominal wall and deeper, organ-related pain. The main goal is to see if there's a difference in pain at rest six hours after surgery. The study will also look at pain at later time points, the amount of opioid medication needed, how quickly women can walk, and when they start breastfeeding.

A total of 156 women will be randomly assigned to receive one of the two blocks after standard spinal anesthesia. Pain will be measured using a simple 0-10 scale at 6, 12, and 24 hours, both at rest and during movement. The study follows strict ethical rules, ensures patient privacy, and all results-whether positive or negative-will be shared to help improve pain management after cesarean delivery.

DETAILED DESCRIPTION:
This study is a prospective, monocentric, randomized controlled trial designed to compare the analgesic efficacy of the transversus abdominis plane (TAP) block versus the erector spinae plane (ESP) block in women undergoing elective cesarean section. Cesarean delivery, one of the most commonly performed surgical procedures worldwide, is associated with both somatic and visceral postoperative pain. Optimizing pain control is critical not only for maternal comfort but also for reducing complications, facilitating early mobilization, and supporting breastfeeding and maternal-infant bonding. While the TAP block provides effective somatic analgesia of the abdominal wall with a rapid learning curve, it does not address visceral pain. Conversely, the ESP block offers multidermatomal coverage, potentially reducing both somatic and visceral components of postoperative pain and opioid consumption. The primary objective of the study is to evaluate postoperative pain at rest six hours after surgery, with secondary outcomes including pain at various time points, opioid consumption, time to first rescue analgesia, ambulation, and initiation of breastfeeding.

A total of 156 patients meeting inclusion criteria (age 18-45 years, elective cesarean, informed consent) will be randomized to receive either a bilateral TAP or ESP block following standardized spinal anesthesia. Pain scores will be assessed using an 11-point Numeric Rating Scale (NRS) at 6, 12, and 24 hours postoperatively, both at rest and with movement. Opioid use, time to ambulation, and breastfeeding initiation will also be recorded. The study is powered to detect a clinically significant difference in pain scores, and data analysis will include tests for normality, parametric and non-parametric comparisons, repeated-measures analysis, regression models, and survival analysis for time-to-event outcomes. The trial adheres to ethical standards, including informed consent and data privacy, and the results will be disseminated regardless of outcome, contributing to evidence-based practice in post-cesarean analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Elective cesarean section
* Ability to provide informed consent

Exclusion Criteria:

* Allergy to any of the drugs used in the study
* Heart disease with impaired cardiac function
* Stage III or higher kidney failure
* Coagulation disorders (platelets <100,000/μL or INR >1.5) or severe liver disease
* Degenerative central nervous system diseases or peripheral neuropathies
* Previous uterine surgery (e.g., myomectomy)
* Previous cesarean section

Pre-pregnancy weight <55 kg

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Pain at Rest at 6 hours | 6 hours after end of surgery
  Pain measured at Rest with Numeric Rating Scale (minimun 0- maximum 10) with 0 meaning no pain and 10 high pain

SECONDARY OUTCOMES:
Pain at Rest at 12 hours | 12 hours after end of surgery
  Pain measured at Rest with Numeric Rating Scale (minimun 0- maximum 10) with 0 meaning no pain and 10 high pain
Pain at Rest at 24 hours | 24 hours after end of surgery
  Pain measured at Rest with Numeric Rating Scale (minimun 0- maximum 10) with 0 meaning no pain and 10 high pain
Pain at Movement at 6 hours | 6 hours after end of surgery
  Pain measured at Rest with Numeric Rating Scale (minimun 0- maximum 10) with 0 meaning no pain and 10 high pain
Pain at Movement at 12 hours | 12 hours after end of surgery
  Pain measured at Rest with Numeric Rating Scale (minimun 0- maximum 10) with 0 meaning no pain and 10 high pain
Pain at Movement at 24 hours | 24 hours after end of surgery
  Pain measured at Rest with Numeric Rating Scale (minimun 0- maximum 10) with 0 meaning no pain and 10 high pain
Milligram of Morphine equivalents in the first 24 postoperative hours | from the end of the surgery to 24 hours after the surgery
  Milligram of Morphine equivalents administered in the first 24 hours
Time to rescue analgesic requirement | Form the end of the surgery to the first rescue analgesic requirement (up to o 24 hours after the surgery)
  Time the patients will require the first rescue analgesic requirement measured in minutes
Time to breast feeding | Form the end of the surgery to the start of breast feeding (up to o 24 hours after the surgery)
  Time the patients will breast feed expressed in minutes
Time to deambulate | Form the end of the surgery to the start of deambulation (up to o 24 hours after the surgery)
  Time the patients will deambulate expressed in minutes

IPD SHARING:
Plan to Share IPD: Undecided